CLINICAL TRIAL: NCT05650762
Title: Controlling Malodour In Fungating Wounds Using A Cinnamon-Based Dressing: Observational Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CEMAG Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIN-S22001
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Wound
Keywords: Malodorous wound; Quality of life; Patient and Investigator discomfort
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cinnamon (Experimental)
  Interventions: Device: Cinesteam

INTERVENTIONS:
Device: Cinesteam — Cinnamon-based Secondary dressing

SUMMARY:
The purpose of the study is to observe the contribution of the cinnamon dressing to the reduction of the discomfort associated with the odour felt by the patient and carers.

This prospective study aims to collect data on patients living with a malodorous fungating wound. Quality of life tools will be used to assess the impact of the cinnamon dressing on managing malodorous fungating wounds.

DETAILED DESCRIPTION:
There are several anti-odour treatments on the market for managing malodorous wounds but no conclusive data on their efficacy is available. Current treatments like charcoal dressing or topical antimicrobials do not completely manage bad odours in particular for tumoral wounds. In the case of malodorous wounds, the ideal management plan would therefore be to reduce (or neutralise) bad odours, and modify any residual odour so that it becomes more pleasant than unpleasant.

Cinesteam® was specially developed to reduce and manage malodorous wounds. Cinesteam® is a secondary dressing that eliminates unpleasant odours and masks any residual odours with the spice's natural fragrance. This dressing also absorbs excess exudates released by the wound.

The aim of this post-market observational study is to observe the performance of Cinesteam® in controlling malodour in fungating wounds. Patients with malodourous, fungating wounds, above 18 years with a discomfort score of >40/100, with cognitive ability to participate and consent, will be eligible to participate in the study. The study will be conducted on eligible patients in the North East of England, treated at the Newcastle upon Tyne Hospitals NHS Foundation Trust, either as inpatients or in its surrounding community.

The duration of patient participation in the study is 14 days. The research nurse will visit patients on Day0 and perform wound assessment, apply Cinesteam dressing over the standard care primary dressing and answer questionnaires on odour, and discomfort, and also help patients with questionnaires on odour, discomfort, appetite and Quality of life.

The research nurse will change Cinesteam dressing on Day 1, Day 7 +/- 48 hours, and Day 14 +/- 48 hours and perform follow-up assessments on patients' wound condition. Patients or their caregivers who usually change the patient's dressing will change the primary dressing and Cinesteam dressing in-between the research nurse's assessment visits. They will keep a record of these dressing changes in the diary provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old with malodorous fungating wounds
* Discomfort > 40/100 expressed by the patient);
* Patients who have capacity to consent;
* Patients who are cognitively able and willing to participate;
* Patients who have a good command of the English language.

Exclusion Criteria:

* Patient with pressure ulcers, leg ulcers, diabetic feet ulcers;
* Terminally ill patients whose life expectancy is less than the duration of the protocol;
* Patients having had metronidazole treatment for fewer than 3 days before enrolment in the study;
* Patients who are unable or willing to participate;
* Anosmic patient (with no sense of smell);
* Patient with cinnamon allergy;
* Persons deprived of their liberty or under guardianship;
* Unable to take part in study procedures for whatever reason;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline patient wound odour at different timepoints using a Visual Analogue Scale (VAS-100mm scale), from 0 (no smell) to 100 (worst smell imaginable) | Baseline visit, one day, 7 and 14 days after baseline visit

SECONDARY OUTCOMES:
Change from baseline patient discomfort associated with the wound odour at different timepoints using a Visual Analogue Scale (VAS-100mm scale), from 0 (no discomfort) to 100 (Unbearable discomfort during the sleeping and waking hours) | Baseline visit, one day, 7 and 14 days after baseline visit
Change from baseline patient quality of life at different timepoints using the questionnaire of EuroQol 5 Dimension 5 Level (EQ-5D-5L) | Baseline visit, one day and 14 days after baseline visit
Change from baseline investigator-rating the strength of the wound odour and smell at different timepoints using TELERTM from none odour to very strong odour. | Baseline visit, one day, 7 and 14 days after baseline visit

CONTACTS AND LOCATIONS:
Locations (1):
- The Newcastle upon Tyne Hospital NHS Foundation Trust, Newcastle upon Tyne, United Kingdom